CLINICAL TRIAL: NCT07221383
Title: A Pilot Randomized Controlled Trial of LDART, a Social Support Intervention for Alcohol Use Disorder
Brief Title: LDART for Alcohol Use Disorder
Acronym: LDART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000040798; K12DA000167 (NIH)
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder; Hazardous Alcohol Use
Keywords: social support; digital intervention; mutual-help groups; alcohol use disorder; addiction recovery
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDART (Experimental): Participants will be given access to LDART for 28 days.
  Interventions: Behavioral: LDART; Behavioral: Resource list
- Resource list (Other): Participants will be emailed a 3-page resource list.
  Interventions: Behavioral: Resource list

INTERVENTIONS:
Behavioral: LDART — Let's Do Addiction Recovery Together! (LDART) is a web-based intervention designed to be used for a few minutes each night to reduce hazardous alcohol use. It has three active ingredients: 1) daily recovery goal setting and tracking, 2) motivational video, audio, and written messages from individuals in recovery, and 3) information on several community-based addiction recovery groups (e.g., support groups).
  Arms: LDART
Behavioral: Resource list — This is a 3-page list of community-based addiction recovery groups that will be emailed to participants. This list was created by the Substance Abuse and Mental Health Services Administration (SAMHSA).

SUMMARY:
This study is a pilot randomized controlled trial to evaluate feasibility, acceptability, and preliminary efficacy of a digital intervention called Let's Do Addiction Recovery Together! (LDART) in adults with alcohol use disorder, relative to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Currently reside in Connecticut, USA
* Have a smartphone that can send and receive text messages and have internet access that can be access over the course of a month
* Had ≥5 heavy drinking days (defined as ≥4 or ≥5 drinks in one sitting for women and men, respectively) in the past 28 days
* AUDIT score of ≥15, indicating moderate/severe AUD
* Alcohol Symptom Checklist ≥4, indicating moderate/severe AUD
* Have some self-reported desire to cut down or quit drinking

Exclusion Criteria:

* Unable to provide informed consent, as assessed by the consent quiz
* Unable to speak, read, or write in English
* Vulnerable population status
* Unlikely to be able to complete study procedures in the next 2-3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From enrollment to the final assessment time point (Day 56)
  The percentage of eligible participants who are enrolled relative to the total number of eligible potential participants who completed the screening.
Accrual rate | From enrollment to the final assessment time point (Day 56)
  The rate of enrollment, defined as number of participants enrolled per month.
Retention rate | From enrollment to the final assessment time point (Day 56)
  The percentage of enrolled participants who complete study-related procedures (i.e., assessment #3).
Intervention engagement | From beginning the intervention (Day 1) to the end of the intervention period (Day 28)
  Number of nights that participants in the active condition completed the activities on the LDART website, out of 28 nights.
Intervention acceptability | The second assessment time point (post-intervention, Day 28)
  Rating scores on the end-user version of the Mobile App Rating Scale (uMARS). Total score range 1-5 with higher scores indicating a better quality app.

SECONDARY OUTCOMES:
Change from baseline in number of drinking days | Baseline (Day 0), Post-intervention (Day 28), 1-month post-intervention (Day 56)
  Change in self-reported number of drinking days in the past 28 days, as measured using the Timeline Follow-back.
Change from baseline in number of heavy drinking days | Baseline (Day 0), Post-intervention (Day 28), 1-month post-intervention (Day 56)
  Change in self-reported number of heavy drinking days (defined as 4 or more drinks for women or 5 or more drinks for in one sitting) in the past 28 days, as measured using the Timeline Follow-back.
Change from baseline in number of recovery groups engaged with | Baseline (Day 0), Post-intervention (Day 28), 1-month post-intervention (Day 56)
  Self-reported number of recovery groups engaged with in the past 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Li Yan McCurdy, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No